CLINICAL TRIAL: NCT03636555
Title: Intranasal Oxytocin Treatment for Alcohol Use Disorders: A Randomized, Placebo-Controlled Trial
Brief Title: Oxytocin Treatment for Alcohol Use Disorders
Acronym: OT-ETOH-4
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI no longer employed at Institution
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-1758; R01AA025942-01A1 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Use Disorder
Keywords: Oxytocin; Heavy drinking; Moderate drinking
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: UNC Hospitals Investigational Drug Service blind labels intranasal spray bottles containing oxytocin or placebo spray and dispenses bottles based on a randomization scheme provided by the study Biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Syntocinon Spray (intranasal oxytocin spray). Each dose is 10 intranasal insufflations totaling 1.0 mL of Syntocinon Spray containing 40 IU of oxytocin. Subjects self-administer doses twice daily (before breakfast and before dinner) for 12 consecutive weeks.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Each dose is 10 intranasal insufflations totaling 1.0 mL of a solution containing all ingredients in Syntocinon Spray except oxytocin. Subjects self-administer doses twice daily (before breakfast and before dinner) for 12 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin will be given in an intranasal spray (Syntocinon Spray) twice daily (10 insufflations, 1.0 mL, 40 IU/dose) for 12 weeks
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Placebo solution (contained all the ingredients in Syntocinon Spray except for oxytocin) will be given as an intranasal spray twice daily (10 insufflations, 1.0 mL/dose) for 12 weeks
  Arms: Placebo

SUMMARY:
To further test the effectiveness of oxytocin in heavy drinkers, half of the cohort in the proposed study will meet criteria for heavy drinking (>35 standard drinks/week [men], >28 standard drinks/week [women] for at least 4 consecutive weeks). However, the investigators think it important to expand the cohort of the proposed study to include subjects with moderate Alcohol Use Disorder (AUD) who meet lower drinking criteria so the outcome of the study will be relevant to a larger percentage of individuals who have AUD. The lower drinking criteria will be minimum of 14 drinks/week (women) or 21 drinks/week (men) with an average of at least two heavy drinking days (≥5 standard drinks for men and ≥4 standard drinks for women) each week in the 4-week period prior to screening. As in the R21-funded Preliminary Study, individuals recruited from the community who meet study criteria based on assessment during a screening clinic visit will be randomized to twice a day (BID) intranasal oxytocin or intranasal placebo during a subsequent clinic visit. After instruction by research staff during the randomization clinic visit, subjects will self-administer intranasal treatments from blind-labeled spray bottles that they take home. During clinic visits at 1, 2, 3, 4, 6, 8, 10, and 12 weeks after randomization, drinking since the last visit will be quantified and other measures summarized above will be obtained. Subjects will self-administer test intranasal treatments for 12 weeks. Drinking will also be quantified during clinic visits at 6 and 12 weeks after cessation of intranasal treatments.

This clinical trial will be the first adequately powered, double blind, placebo-controlled trial examining the efficacy and tolerability of BID intranasal oxytocin (40 IU/dose; 80 IU/d) on alcohol drinking in AUD. The trial will also be the first to prospectively examine the effects of intranasal oxytocin on anxiety symptoms in individuals with AUD.

DETAILED DESCRIPTION:
Design: This will be a randomized, double blind, 12-week clinical trial comparing the efficacy of intranasal self-administration of oxytocin (Syntocinon Spray [intranasal oxytocin spray], Novartis) vs. intranasal placebo (containing the same ingredients as Syntocinon Spray except for oxytocin) to in individuals with moderate Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) AUD and individuals with severe AUD who, in both groups, meet specific drinking criteria. Treatment assignments will be counterbalance within gender and within the moderate and severe AUD groups. The primary outcomes are measures of drinking: percentage of heavy drinking days (>5 [men], >4 [women] standard drinks), percentage of abstinent days, and mean standard drinks per drinking day based on Timeline Followback interview data collected at each clinic visit after randomization (1, 2, 3, 4, 6, 8, 10, and 12 weeks during the intranasal test treatment period; 6 and 12 weeks after cessation of test treatments). Secondary outcomes are subject self-ratings of craving for alcohol and anxiety on standardized questionnaires. Baseline measures of drinking, craving and anxiety will be covariates in statistical comparisons between the treatment groups of outcomes over the course of the treatment trial and the follow-up period.

Procedures Recruitment: Potential participants will be recruited from the Raleigh, Durham, and Chapel Hill, North Carolina areas by screening subjects who respond to community advertising. Respondents to advertisements will have a preliminary telephone screening conducted by the study coordinator. Individuals who appear eligible, as determined by the investigative team, will be scheduled for more comprehensive in-person screening.

Screening Clinic Visit: Prospective subjects who appear to meet study criteria based on phone interviews will come to the Psychiatry outpatient clinic at a scheduled time for in-person screening procedures to ascertain whether they truly meet study criteria (see Eligibility Criteria below). Initially individuals will read and sign the informed consent and be given a copy for their records. A breathalyzer test using an Alco-Sensor III breathalyzer machine (Intoximeters, Inc., St. Louis, MO) will be administered [breath alcohol concentration (BrAC) must be 0.00 gms/dL to give informed consent]. Medical personnel will administer the Clinical Institute Withdrawal Assessment of Alcohol (CIWA) Scale to determine if subjects are exhibiting significant alcohol withdrawal. The CIWA score must be <6 for subjects to give informed consent. If the score is >6, the visit will be rescheduled. In addition, blood pressure (BP) and heart rate (HR), height and weight will be measured and BMI calculated. Medical personnel will conduct a medical history and examination including a neurological examination. Over-the-counter and prescription medication use will be recorded. The Fagerstrom Test for Nicotine Dependence will be administered to smokers. Laboratory evaluations will include complete blood count (CBC) with differential; chemistries including bilirubin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Gamma-glutamyl transferase (GGT), sodium, potassium, chloride, blood urea nitrogen, creatinine, and glucose; and urinalysis as well as urine toxicology (drug screen). A carbohydrate deficient transferrin (CDT) sample will be drawn. CDT samples will be stored frozen and then shipped in batches of 40 to Dr. Ray Anton's lab in Charleston, South Carolina for assay. CDT demonstrates excellent specificity to detect heavy alcohol use over time and has been shown to complement self-report measures of consumption. With subjects' permission, a sample of blood will also be obtained to archive for possible future genetic analyses. Women will be given a serum pregnancy test (β-HCG) at screening and a urine pregnancy test at wks 4, 8, and 12. Trained interviewers will conduct the psychiatric/substance disorder-screening interview using the Mini International Neuropsychiatric Interview. The Structured Clinical Interview for DSM-V Substance Use Disorders Module for AUD will be completed by a study physician to determine criteria for moderate or severe AUD. The study coordinator will conduct the pretreatment 90-day Timeline Followback interview (TLFB, Sobell et al, 1988) and potential participants will complete the entire Spielberger State Trait Anxiety Inventory (SSTAI), the Drinker's Inventory of Consequences, the Family History of Alcoholism Module (FHAM) to assess family history of alcohol problems, the University of Rhode Island Change Assessment Scale to assess motivation level, the Penn Alcohol Craving Scale to assess baseline craving, and the Insomnia Severity Index to assess baseline sleep problems. Additionally, potential participants will fill out a short evaluation of their treatment goals. This visit should take about 3 h.

Randomization Clinic Visit: Individuals meeting inclusion but not exclusion criteria will be informed and scheduled for the initial treatment visit within 10 days. Eligible individuals will not be required to abstain from drinking alcohol prior to randomization. The study coordinator will administer a breathalyzer test (BrAC must be ≤0.04 gm/dL; if >0.04 gm/dL, the visit will be rescheduled), measure BP and HR, conduct the TLFB interview, and ask participants to complete the PACS, the state portion of the SSTAI (SSAI), and the Fagerstrom Test. After BrAC reading, but before the other procedures, the study physician will evaluate withdrawal symptoms using the CIWA and note the use of medications. If the CIWA score is >6, the visit will be rescheduled. A 60 mL bottle containing 50 mL of test substance (oxytocin or placebo solution) with an intranasal spray mechanism that ejects 0.1 mL of aerosolized solution per insufflation as well as written instructions will be dispensed from the UNC Hospitals Investigational Drug Service according to the randomization schedule provide by Dr. Robert Gallop, Biostatistical Consultant on the project. The bottle will contain sufficient solution for the subject to self-administer intranasal test substance for at least 18 days so he/she will not run out if there is a delay in returning for the next clinic visit. Subjects will receive instructions for self-administration of intranasal test substance from members of the Study Team. Subjects will then self-administer their first dose of the intranasal substance to which they have been randomized [ten insufflations delivering 40 IU of Syntocinon (oxytocin) Spray in a total of 1.0 mL of solution, or the same volume of placebo solution which contains all the ingredients in Syntocinon Spray except oxytocin]. Subjects will pause 30 sec between insufflations and will alternate insufflations between nostrils. Study Team members will observe subjects' self-administration of their first dose to determine if their technique is correct and to correct any errors in technique. In our experience, subjects rapidly learn the self-administration technique. Participants also will be given a calendar style diary to record times of intranasal self-administration, drinking, and any side effects and a Self-Administration Instruction Sheet along with a wallet card informing providers that the subject may be taking oxytocin should the individual require emergency medical treatment. Finally, participants will receive Medical Management (MM) from a trained clinician (see details below). This visit should be completed in about 1.25-1.5 hours.

Subsequent Clinic Visits: Subjects will self-administer intranasal test doses BID (before breakfast and dinner) for 12 weeks. They will have outpatient clinic visits at weeks 1, 2, 3, 4, 6, 8, 10 and 12 after starting intranasal test treatments. The investigators will accept a window of ± 3 days for weekly visits and ± 7 days for biweekly visits in cases where a subject cannot come for the exact visit date. At each visit, the following will be obtained: breathalyzer (BrAC) reading; CIWA score; TLFB interview; BP; HR; the state portion of the SSTAI; and PACS. The DrInC will be completed again at week 12. BrAC readings must be <0.04 and CIWA scores <6 for assessments to be done at clinic visits (BrAC readings must be <.08 to allow subjects to drive themselves home from any clinic visit). New spray bottles will be given every 2 weeks. The weight of bottles will be recorded when first issued and when returned during subsequent clinic visits. Change in weight will be our primary measure of compliance. Blood and urine samples will be obtained for CBC, electrolytes, Blood Urea Nitrogen (BUN), creatinine, liver function tests, urinalysis, urine drug screen and pregnancy tests at 4, 8, and 12 weeks. As during the randomization clinic visit, the psychosocial treatment provided during each subsequent clinic visit will be Medical Management (MM). At the 12-week clinic visit, subjects will be given information about a wide range of treatment options as well as contact information and will be offered assistance in making appointments.

Post-Treatment Follow-up: Subjects will return for follow-up clinic visits at 6 and 12 weeks (2 weeks also for follow-up measures if lab values at the 12-week clinic visit during the test treatment period are abnormal) after cessation of intranasal test treatments. Assessment at each follow-up visit will be BrAC, TLFB, PACS, SSAI, and questions about subjects' enrollment and attendance record in individual, group, and/or medication treatment.

Medical Management Intervention: The psychosocial treatment for the proposed study will be Medical Management (MM). Dr. Kampov will be primarily responsible for MM with Drs. Garbutt, Jordan and Pedersen providing additional coverage. Dr. Kampov and Dr. Garbutt have been trained and certified in MM by Dr. William Dundon of the University of Pennsylvania and along with Drs. Pedersen and Jordan have received MM training from Ms. Gail Kempf of the University of Pennsylvania. MM is designed as a means for physicians and other health care providers to encourage individuals with an AUD to make progress towards their drinking goals of reduction or abstinence and to encourage compliance with medication. Whereas the primary goal of MM is to encourage abstinence, the goal of reduction is acceptable and the investigators have used this "harm reduction" approach in our clinical trials to date. Many subjects have an initial goal of reduction that, over the course of trial participation, MM changes to abstinence. MM does not provide intense counseling methods for reducing drinking or dealing with relapse triggers and is thought to be an advantage for medication trials as MM does not overpower a possible medication effect. The average length of MM sessions is 10-15 minutes and an MM checklist is used in each session that greatly enhances consistency. The investigators will audio-record 10-20 MM sessions for review by MM providers to enhance fidelity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 21 and 65. Children, ages less than 21 years, and adults over 65 years will not be studied because of the lack of safety data on the use of oxytocin in these age ranges.
2. All subjects must meet DSM-V criteria for moderate or severe alcohol use disorder. In addition the investigators will recruit 50% of individuals (evenly distributed between men and women) who meet criteria for heavy drinking: > 28 standard drinks/week (women) or >35 drinks/week (men) in the 30-day period prior to screening. Those not meeting heavy drinking criteria will be required to have a minimum of 14 drinks/week (women) or 21 drinks/week (men) with an average of at least two heavy drinking days (≥5 standard drinks for men and ≥4 standard drinks for women) per week in the 30 day period prior to screening
3. Ability to understand and sign written informed consent.
4. Must have a 0.0 gms/dL breathalyzer reading on the day of screening and < 0.4 gms/dL on the day of randomization.
5. Express a desire to achieve abstinence or to greatly reduce alcohol consumption
6. Must have a stable residence and be able to identify an individual who could contact participant if needed.

Exclusion Criteria:

1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., cirrhosis, unstable hypertension, unstable diabetes mellitus). Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, severe depression, or suicidal ideation.
2. Substance use disorder other than nicotine use disorder or mild cannabis use disorder. Occasional use of cocaine is acceptable.
3. Concurrent use of any psychotropic medication including, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics with the exception of stable doses of antidepressants for one month.
4. Prior history of adverse reaction to oxytocin.
5. Serum sodium concentration < 134 mEq/L.
6. Creatinine level > 1.5 times Upper Limit of Normal (ULN) or Estimated Glomerular Filtration Rate < 50.
7. AST, or ALT > 5 times ULN or bilirubin > 1.5 X ULN.
8. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of moderate/severe cannabis use disorder.
9. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
10. Women who are breastfeeding.
11. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol dependence.
12. Participation in any clinical trial within the past 60 days.
13. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Mean heavy drinking days | 24 weeks
  A heavy drinking day is defined by consumption of 5 (men) or 4 (women) standard drinks or more during a day
Mean drinks per drinking day | 24 weeks
  The average number of standard drinks consumed on days when subjects drink alcohol drinks

CONTACTS AND LOCATIONS:
Overall Officials: Cort Pedersen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Cort Pedersen, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Supporting Information: Study Protocol, CSR
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Anton RF. Carbohydrate-deficient transferrin for detection and monitoring of sustained heavy drinking. What have we learned? Where do we go from here? Alcohol. 2001 Nov;25(3):185-8. doi: 10.1016/s0741-8329(01)00165-3. PMID 11839464
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL (2016) Structured Clinical Interview for DSM-5 Disorders-Clinician Version (SCID-5-CV). American Psychiatric Association.
- [Background] Sheehan D, Janavs J, Baker R, Harnett-Sheehan K, Knapp E, Sheenan M (1999) Mini International Neuropsychiatric Interview (M.I.N.I.). Tampa: University of South Florida.
- [Background] Spielberger CD, Gorsuch RL, Lushene RE (1969) The state trait anxiety inventory manual. Palo Alto: Consulting Psychologists Press
- [Background] McConnaughy DA, DiClemente CC, Prochaska JO, Velicer WF (1989). Stages of change in psychotherapy: a follow-up report. Psychother Theory Res Pract 4: 494-503
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Pettinati HM, Weiss RD, Dundon W, Miller WR, Donovan D, Ernst DB, Rounsaville BJ. A structured approach to medical management: a psychosocial intervention to support pharmacotherapy in the treatment of alcohol dependence. J Stud Alcohol Suppl. 2005 Jul;(15):170-8; discussion 168-9. doi: 10.15288/jsas.2005.s15.170. PMID 16223068
- [Background] Miller WR, Tonigan JS, Longabaugh R (1995) The Drinker Inventory of Consequences (DrInC): An instrument for assessing adverse consequences of alcohol abuse. Project MATCH Monograph Series, Vol. 4. Rockville, MD: NIAAA
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Rice JP, Reich T, Bucholz KK, Neuman RJ, Fishman R, Rochberg N, Hesselbrock VM, Nurnberger JI Jr, Schuckit MA, Begleiter H. Comparison of direct interview and family history diagnoses of alcohol dependence. Alcohol Clin Exp Res. 1995 Aug;19(4):1018-23. doi: 10.1111/j.1530-0277.1995.tb00983.x. PMID 7485811